CLINICAL TRIAL: NCT04678778
Title: Targeted Physical and Cognitive Activity in a VR Environment - COVID-19 Protocol
Brief Title: Virtual Reality Study - COVID-19 Protocol
Acronym: NRVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Judy Pa, Associate Professor of Neurology, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS17-00354
Record Dates: First submitted 2020-12-11; First posted 2020-12-22 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Healthy Aging
Keywords: Virtual Reality; VR; Cognitive Activity; Physical Activity; Bike; Cycling; Intervention; USC; Brain Health
MeSH Terms: conditions — Motor Activity | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined, simultaneous physical and cognitive activity (Experimental): The combined physical and cognitive activity VR arm will participate in our customized spatial navigation program that increases difficulty and length per trial over time. As described in the Game Design section, each session will consist of 5 trials. The first trial will be a long-delay free recall condition from the previous day's path. The next 4 trials will consist of learning, cued recall, and free recall. This VR-based spatial navigation program has been tested in our feasibility trial for safety and tolerability in older adults.
  Interventions: Behavioral: Physical and Cognitive Activity

INTERVENTIONS:
Behavioral: Physical and Cognitive Activity — There are three sessions a week for the course of 12 weeks. Each session consists of 5 trials.

SUMMARY:
The overarching goal of this pilot clinical trial is to use a novel virtual reality (VR)-based intervention that simultaneously engages physical and cognitive activity aimed at improving brain and cognitive outcomes in older adults. Physical activity is a promising lifestyle intervention for mitigating cognitive decline or delaying onset of dementia. However, to fully leverage beneficial brain effects of physical activity, training the brain to learn and engage in a cognitively stimulating environment may be the key to enhanced brain and cognitive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 50-85 Years Old
* Able to Walk Without Assistance
* Fluent in English
* No Ferromagnetic Metal in Body
* Able to Participate in Moderate Aerobic Physical Activity

Exclusion Criteria:

* Severe Brain Injury/ Head Trauma
* Pacemakers or Metal Implants
* Claustrophobia
* Contradictions to Magnetic Resonance Imaging (MRI)/ Positron Emission Tomography (PET) Brain Scans
* Opposition to Blood Draws

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Image (MRI) brain scan of hippocampal volume (cubic mm) | 12 weeks
  The hippocampus has been shown to be a selectively vulnerable region in Alzheimer's Disease (AD), and several studies, including our own, identified a dysfunctional brain signal in the hippocampus in Mild Cognitive Impairment (MCI) patients. We propose to examine the effects of exercise on remediating this hyperactive signal exhibited in MCI patients.
Mnemonic Similarity Task for visual memory performance - discrimination index | 12 weeks
  With the study's primary focus on hippocampal function, we will use the Mnemonic Separation Task (MST), a hippocampus-dependent discrimination test of similar objects, as our primary cognitive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Pa, PhD, Principal Investigator — University of Southern California
Locations (1):
- Mark and Mary Stevens Neuroimaging and Informatics Institute of the University of Southern California, Los Angeles, California, United States